CLINICAL TRIAL: NCT00835939
Title: Treatment for Achilles Tendinopathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Sport Science Association of Alberta (SSAA) (Unknown)
Responsible Party: Dr. J Preston Wiley, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UC-20903-RR
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Achilles Tendinopathy; Achilles Tendon Enthesopathy; Mid-Portion Achilles Tendinopathy; Insertional Achilles Tendinopathy; Non-Insertional Achilles Tendinopathy
Keywords: Achilles; Tendinopathy; Sclerotherapy; Neovascularisation; sports medicine; interventional radiology
MeSH Terms: conditions — Tendinopathy; Neovascularization, Pathologic | interventions — Glucose; Lidocaine; Sclerotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25% Dextrose and 1% Lidocaine (Active Comparator)
  Interventions: Drug: 25% Dextrose and 1% Lidocaine; Procedure: sclerotherapy
- Lidocaine (Placebo Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: 25% Dextrose and 1% Lidocaine — Up to 3 injections provided to neovessels outside of the tendon
  Arms: 25% Dextrose and 1% Lidocaine
Drug: Lidocaine — Up to 3 injections provided to neovessels outside of the tendon
  Arms: Lidocaine
Procedure: sclerotherapy
  Arms: 25% Dextrose and 1% Lidocaine

SUMMARY:
The purpose of this study is to determine whether sclerotherapy using a 25% dextrose and 1% lidocaine solution is an efficacious treatment for patients with chronic Achilles tendinopathy who have failed a home based, heavy load eccentric training program.

DETAILED DESCRIPTION:
The purpose of this research project is to optimize the clinical outcome of patients with Achilles tendinopathy. Patients who fail a standardized physical therapy regiment (eccentric training protocol) will be randomly allocated into two groups with one group receiving an injection of hypertonic glucose and Lidocaine (sclerosing solution) and the other receiving an injection of Lidocaine (control). Neovascularisation (growth of new blood vessels and nerves into a damaged area of the tendon) appears to be associated with pain and subsequently a decrease in function and use of the affected tendon. Results of an observational study in Sweden revealed that in all patients for which eccentric training was unsuccessful neovascularisation was present. Sclerosis of neovessels appears to be successful in removing the pain associated with Achilles tendinopathy in both mid-portion and enthesitis patients. However, there are no studies that have administered this technique to a homogenous patient population in a prospective, controlled and randomized manner. In addition, there are no studies that have compared the effects of eccentric training in healthy individuals versus patients with painful Achilles tendinopathy in a controlled longitudinal study. It is expected that patients for whom eccentric training is unsuccessful and who subsequently receive sclerosing therapy will show a statistically significant improvement in pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older with a minimum of 3 months of clinically determinant history and symptoms (pain) consistent with unilateral Achilles tendinopathy (enthesitis or mid-portion) as diagnosed by a sport medicine physician.
* Participants are not required to have tried other treatments, however, those who have tried other treatments (except injection treatments) including, but not restricted to, oral NSAIDs, topical NSAIDs, shoe modifications, and physical/athletic therapy will not be restricted from the study
* Provide informed consent for the controlled longitudinal study and RCT

Exclusion Criteria:

* Individuals with physical ailments precluding them from performing the eccentric training program
* Worker's Compensation Board (WCB) and elite athletes (varsity, national and professional level).
* Individuals younger than 18 years of age will be excluded from this trial due to the complicating factors of musculoskeletal immaturity and the lack of relevant research of Achilles tendinopathy and neovascular bundles in this population.
* Previous Achilles tendon rupture of the tendon in question
* Individuals that have received any type of injection in or around the Achilles tendon
* Known allergy to dextrose based sclerosing agent or other contraindications
* Known allergy to Lidocaine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute for Sport Assessment - Achilles | Baseline, 4 weeks, 8 weeks, 12 weeks, 6 months, 1 year

SECONDARY OUTCOMES:
100 mm Visual Analog Scale | Baseline, 4 weeks, 8 weeks, 12 weeks, 6 months, 1 year
Tegner Activity Scale | Baseline, 4 weeks, 8 weeks, 12 weeks, 6 months, 1 year
Number of Neovessels | Baseline, 4 weeks, 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J Preston Wiley, MD, MPE, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada